CLINICAL TRIAL: NCT03119051
Title: Shanghai Non-pharmacological Intervention of Mild Cognitive Impairment for Delaying Progress With Longitudinal Evaluation
Brief Title: Shanghai Non-pharmacological Intervention of Mild Cognitive Impairment
Acronym: SIMPLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Binyin Li, Principle Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuijinHSH
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Dysfunction
Keywords: mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- online cognitive training (Experimental): Patients will receive 3-4 times of 20-30 minutes' training game every week
  Interventions: Behavioral: Online cognitive training
- no training (No Intervention): Patients will not undergo preoperative cognitive training.
- Cognitive training and physical exercise (Experimental): Patients will receive 3-4 times of 20-30 minutes' training game every week and 2 times of 60 minutes' Tai Chi Training
  Interventions: Behavioral: Cognitive training plus physical exercise

INTERVENTIONS:
Behavioral: Online cognitive training — A variety of cognitive domains will be involved in the training including memory, calculation, attention, visuospatial and executive skills. The difficulty level of each game will be adjusted automatically according to patients' last training results so that patients' correction rate will be kept between 70% and 80%.
  Arms: online cognitive training
Behavioral: Cognitive training plus physical exercise — Online cognitive training A variety of cognitive domains will be involved in the training including memory, calculation, attention, visuospatial and executive skills. The difficulty level of each game will be adjusted automatically according to patients' last training results so that patients' correction rate will be kept between 70% and 80%.
  Physical Exercise Tai Chi Training：a teacher will give two 60-min lessons per week. Participants will play Tai Chi in the lessons, following teacher's instruction.
  Arms: Cognitive training and physical exercise

SUMMARY:
This study evaluates the effects of "computerized cognitive training" and "cognitive training plus exercise training" on different cognitive domains in mild cognitive impairment (MCI) patients. Patients will be randomized into the computerized training group, cognitive training plus exercise training group and the control group.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is an early stage of Alzheimer Disease (AD). Increasing evidence has indicated that cognitive trainings improve cognition functions of MCI patients in multiple cognitive domains, making it a promising therapy for MCI. However, the effect of long-time training has not been widely explored. It is also necessary to evaluate the extent of its function in reducing the conversion rate from MCI to AD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 50-85;
* MCI diagnosed according to the National Institute on Aging-Alzheimer's Association (NIA-AA) workgroups[1];
* 24≤Mini-Mental State Examination (MMSE) ≤28；
* The Hamilton Depression Scale/17-item (HAMD) score ≤10;
* Not on medication for dementia;
* MRI T2 weighted image (T2WI) scan: aged ≤70 , Fazeca scale for White Matter lesions rating level≤1; >70 years, white matter damage rating scale ≤2. The number of lacunar infarcts larger than 2 cm in diameter ≤2. No infarcts in hypothalamus, entorhinal cortex, para-hypothalamus, cortical and subcortical cavity infarction near gray matter nuclei. The medial temporal lobe atrophy (MTA) score: Grade II or above.
* Accompanied by reliable caregivers (at least intensive contact of 4 days every week and 2 hours every day) who are expected to participate in the follow-up visits and provide useful information for scores of scales like ADCS-ADL;
* Education level: primary school (grade 6) or above.
* Expected good compliance with the therapy and follow-up. Each patient gives a written informed consent, and the study has been approved by Ruijin Hospital's ethical committees.

Exclusion Criteria:

* Cognitive decline caused by other diseases (cerebrovascular disease, central nervous system infections, Parkinson's disease, metabolic encephalopathy, intracranial space-occupying lesions, deficiency of folic acid/vitamin B12 and hypothyroidism);
* Medical history of other neurological disorders (including stroke, Neuromyelitis optica, Parkinson's disease, epilepsy, etc.);
* Psychiatric disorders defined by (Diagnostic and Statistical Manual of Mental Disorders) DSM-IV criteria;
* Unstable or severe disease of heart, lung, liver, kidney or hematopoietic system;
* History of alcohol or drug abuse;
* Participation in other clinical trial less than 30 days before the screening of this study;
* Inability to complete the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of AD | 12 months
  The 3-year incidence of AD in each group will be compared.

SECONDARY OUTCOMES:
The global cognitive function of MCI patients | 6 months
  Alzheimer disease assessment scale (ADAS-Cog) will be used to assess the global cognitive performance of MCI patients
Memory | 12 months
  Memory will be assessed using the Auditory verbal learning test-Huashan version (AVLT-H).
Attention | 12 months
  Attention will be evaluated by Trial Making Test (TMT).
Executive functions | 12 months
  Executive functions will be evaluated by the Stroop task.
Language | 12 months
  Language will be assessed by Boston naming test (30-item version).
Visual spatial ability and visual memory | 12 months
  Visual spatial ability and visual memory will be evaluated by the Rey-Osterrieth complex figure test (CFT).
Activities of daily living | 6 months
  Activities of daily living will be assessed by Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL).
Structural MRI | 12 months
  Volume of hippocampus and other specific brain regions
Gut microbiota | 12 months
  Number of genera and abundence of E.coli in feces and blood

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Di Chen, Study Director — Rui Jin Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Y, Li B, Tang H, Xu Q, Wu Y, Cheng Q, Li C, Xiao S, Shen L, Tang W, Yu H, He N, Lin H, Yan F, Cao W, Yang S, Liu Y, Zhao W, Lu D, Jiao B, Xiao X, Zhou L, Chen S. Shanghai cognitive intervention of mild cognitive impairment for delaying progress with longitudinal evaluation-a prospective, randomized controlled study (SIMPLE): rationale, design, and methodology. BMC Neurol. 2018 Jul 24;18(1):103. doi: 10.1186/s12883-018-1100-x. PMID 30041656